CLINICAL TRIAL: NCT03315156
Title: Taste Changes in Acute Otitis Media
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: TASMC-17-AD-0311-17-TLV-CTIL
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Acute Otitis Media
Keywords: Acute otitis media; AOM; Electrogustometer; EGM; Taste threshold
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: patients with AOM
  Interventions: Diagnostic Test: Electrogustometery

INTERVENTIONS:
Diagnostic Test: Electrogustometery — Taste assessment using EGM

SUMMARY:
Detection of taste changes in Acute Otitis Media (AOM) patients.

DETAILED DESCRIPTION:
Methods:

Taste assessment will be done using Electrogustometer (EGM). Tongue stimulation will be performed using low currents of up to 100uA. Using the protocol as specified in the EGM user manual.

Population: 40 Unilateral AOM patients, aged 8-40. Without chronic otitis media, pregnancy or impaired judgement.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral AOM

Exclusion Criteria:

* Chronic Otitis Media
* Pregnancy
* Patients with lack of judgment

Ages: 8 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with AOM
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Taste change in AOM | 1 week
  change in taste threshold in AOM patients

CONTACTS AND LOCATIONS:
Overall Officials: Ari DeRowe, MD, Principal Investigator — TLVMC